CLINICAL TRIAL: NCT01951586
Title: A Randomized, Double-blind, Multi-center Phase 2 Trial of Denosumab in Combination With Chemotherapy as First-line Treatment of Metastatic Non-small Cell Lung Cancer
Brief Title: Denosumab in Combination With Chemotherapy as First-line Treatment of Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20120249; 2013-001662-42 (EudraCT Number)
Record Dates: First submitted 2013-09-24; First posted 2013-09-26 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo matching to denosumab by subcutaneous injection once every 4 weeks plus one loading dose on study day 8 in addition to platinum-based standard chemotherapy. Participants with bone metastases also received 4 mg zoledronic acid administered as an IV infusion Q4W or Q3W.
  Interventions: Drug: Zoledronic acid; Drug: Placebo to Denosumab; Drug: Standard Chemotherapy
- Denosumab (Experimental): Participants received 120 mg denosumab by subcutaneous injection once every 4 weeks plus one loading dose on study day 8 in addition to platinum-based standard chemotherapy. Participants with bone metastases also received placebo to zoledronic acid administered as an IV infusion Q4W or Q3W.
  Interventions: Drug: Denosumab; Drug: Standard Chemotherapy; Drug: Placebo to Zoledronic Acid

INTERVENTIONS:
Drug: Denosumab — Administered by subcutaneous injection once every 4 weeks (Q4W) plus one loading dose on study day 8; could be administered as often as every 3 weeks (Q3W) to participants receiving Q3W chemotherapy.
  Other Names: XGEVA
  Arms: Denosumab
Drug: Zoledronic acid — Administered by intravenous infusion in participants with bone metastasis upon investigative site request for IV bone-targeted therapy.
  Other Names: Zometa
  Arms: Placebo
Drug: Placebo to Denosumab — Administered by subcutaneous injection once every 4 weeks (Q4W) plus one loading dose on study day 8; could be administered as often as every 3 weeks (Q3W) to participants receiving Q3W chemotherapy.
  Arms: Placebo
Drug: Standard Chemotherapy — Standard of care chemotherapy consisting of pemetrexed or gemcitabine in combination with cisplatin or carboplatin administered according to local practice.
Drug: Placebo to Zoledronic Acid — Administered by intravenous infusion in participants with bone metastasis upon investigative site request for IV bone-targeted therapy.
  Arms: Denosumab

SUMMARY:
This randomized phase 2 trial is studying the effect of adding denosumab to standard chemotherapy in the treatment of advanced lung cancer.

DETAILED DESCRIPTION:
This is a global randomized double-blind placebo-controlled study in patients with Stage IV untreated non-small cell lung cancer (NSCLC) with or without bone metastasis. Eligible participants are to receive 4 to 6 cycles of a standard of care platinum-doublet chemotherapy regimen. Participants will be randomized in a 2:1 ratio to receive denosumab or matching placebo with the first investigational product dose coinciding with participant's first cycle of chemotherapy and continuing until the primary analysis, unacceptable toxicity, withdrawal of consent, death, or lost to follow-up. Participants who discontinued the investigational product early (ie, before primary analysis) were followed for disease status and survival. The primary analysis took place when 149 events of death had been reported. All participants were followed for 2 years after the last dose of blinded investigational product.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IV non-small cell lung carcinoma (NSCLC), according to 7th Tumor/Node/Metastasis (TNM) classification (cytological specimens obtained by bronchial washing or brushing, or fine-needle aspiration are acceptable)
* Subject has available and has provided consent to release to the sponsor (or designee) a tumor block with confirmed tumor content (or approximately 20 unstained charged slides [a minimum of 7 slides is mandatory]) and the corresponding pathology report
* Planned to receive 4 to 6 cycles of pemetrexed or gemcitabine in combination with cisplatin or carboplatin

  • For subjects to receive pemetrexed, planned to receive vitamin B12 and folate per pemetrexed approved labeling
* Radiographically evaluable (measurable or non-measurable) disease (according to modified Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria
* Other inclusion criteria may apply

Exclusion Criteria:

* Known presence of documented sensitizing epidermal growth factor receptor (EGFR) activating mutation or echinoderm microtubule-associated protein-like 4-anaplastic lymphoma kinase (EML4-ALK) translocation (screening following local standards, but strongly encouraged in non-squamous histology)
* Known brain metastases (systematic screening of patients not mandatory)
* Any prior systemic therapy (before randomization) for the treatment of NSCLC (including chemoradiation), except if for non-metastatic disease and was completed at least 6 months prior to randomization
* Planned to receive bevacizumab
* Significant dental/oral disease, including prior history or current evidence of osteonecrosis/ osteomyelitis of the jaw, or with the following:

  * Active dental or jaw condition which requires oral surgery
  * Non-healed dental/oral surgery
  * Planned invasive dental procedures for the course of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2013-12-31 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (67):
- United States (17):
  - Research Site, Goodyear, Arizona
  - Research Site, Anaheim, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Farmington, Connecticut
  - Research Site, Alexandria, Louisiana
  - Research Site, Brewer, Maine
  - Research Site, Westminster, Maryland
  - Research Site, Fairhaven, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, East Setauket, New York
  - Research Site, Durham, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Nashville, Tennessee
- Australia (6):
  - Research Site, Kogarah, New South Wales
  - Research Site, Wahroonga, New South Wales
  - Research Site, Adelaide, South Australia
  - Research Site, Footscray, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, Wodonga, Victoria
- Canada (6):
  - Research Site, Edmonton, Alberta
  - Research Site, Saint John, New Brunswick
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Czechia (5):
  - Research Site, Chomutov
  - Research Site, Ostrava-Poruba
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Ústí nad Labem
- France (8):
  - Research Site, Caen
  - Research Site, Dijon
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Reims
  - Research Site, Saint-Quentin
  - Research Site, Tours
- Germany (4):
  - Research Site, Berlin
  - Research Site, Großhansdorf
  - Research Site, Köln-Merheim
  - Research Site, Ulm
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Italy (5):
  - Research Site, Monza (MB)
  - Research Site, Orbassano (TO)
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Saronno VA
- Netherlands (5):
  - Research Site, 's-Hertogenbosch
  - Research Site, Arnhem
  - Research Site, Harderwijk
  - Research Site, Tilburg
  - Research Site, Zutphen
- United Kingdom (7):
  - Research Site, Bristol
  - Research Site, Exeter
  - Research Site, Glasgow
  - Research Site, Guildford
  - Research Site, London
  - Research Site, Plymouth
  - Research Site, Preston

REFERENCES:
- [Background] Peters S, Danson S, Ejedepang D, Dafni U, Hasan B, Radcliffe HS, Bustin F, Crequit J, Coate L, Guillot M, Surmont V, Rauch D, Rudzki J, O'Mahony D, Barneto Aranda I, Scherz A, Tsourti Z, Roschitzki-Voser H, Pochesci A, Demonty G, Stahel RA, O'Brien M. Combined, patient-level, analysis of two randomised trials evaluating the addition of denosumab to standard first-line chemotherapy in advanced NSCLC - The ETOP/EORTC SPLENDOUR and AMGEN-249 trials. Lung Cancer. 2021 Nov;161:76-85. doi: 10.1016/j.lungcan.2021.09.002. Epub 2021 Sep 9. PMID 34543941
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 57 centers in 10 countries including the United Kingdom, Netherlands, France, Italy, Germany, Czech Republic, United States, Canada, Australia and Greece. Participants were enrolled from 31 December 2013 to 21 May 2015.
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive denosumab or placebo. Randomization was stratified based on the presence of bone metastasis (yes or no), histology (squamous versus non-squamous), and geographic region (North America, Western Europe/Australia, and rest of world [ROW]).
Groups:
- Placebo: Participants were randomized to receive placebo matching to denosumab by subcutaneous injection once every 4 weeks (Q4W) plus one loading dose on study day 8 in addition to platinum-based standard chemotherapy. Participants may have received placebo as often as once every 3 weeks (Q3W) while receiving Q3W chemotherapy. Participants with bone metastases also received 4 mg zoledronic acid administered as an IV infusion Q4W or Q3W.
- Denosumab: Participants were randomized to receive 120 mg denosumab by subcutaneous injection once every 4 weeks plus one loading dose on study day 8 in addition to platinum-based standard chemotherapy. Participants may have received denosumab as often as Q3W while receiving Q3W chemotherapy. Participants with bone metastases also received placebo to zoledronic acid administered as an IV infusion Q4W or Q3W.
Period: Overall Study
Arm/Group | Placebo | Denosumab
Started | 78 | 148
Received Study Drug | 76 | 145
Completed | 0 | 0
Not Completed | 78 | 148
Not completed — Death | 61 | 120
Not completed — Withdrawal by Subject | 8 | 17
Not completed — Lost to Follow-up | 0 | 1
Not completed — Sponsor Decision | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Denosumab | Total
Number analyzed (Participants) | 78 | 148 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (10.1) | 63.8 (9.7) | 63.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 54 | 74
  Male | 58 | 94 | 152
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 7 | 9
  White or Caucasian | 73 | 133 | 206
  Others | 3 | 8 | 11
Presence of Bone Metastasis [Count of Participants; unit: Participants] — Data are based on randomized strata.
  Participants
    Yes | 35 | 65 | 100
    No | 43 | 83 | 126
Histology [Count of Participants; unit: Participants] — Data are based on randomized strata.
  Participants
    Squamous | 18 | 35 | 53
    Non-squamous | 60 | 113 | 173
Geographic region [Count of Participants; unit: Participants]
  North America/Australia | 30 | 63 | 93
  Western Europe | 35 | 67 | 102
  Rest of World | 13 | 18 | 31
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participants disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active; 1
  = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self- Care; 4 = Completely Disabled, no self-care, confined to bed or chair; 5 = Dead.
  Participants
    0 (Fully active) | 33 | 69 | 102
    1 (Restrictive but ambulatory) | 45 | 79 | 124
Time from Initial Diagnosis of NSCLC to Randomization [Mean (Standard Deviation); unit: months] | 2.46 (5.28) | 6.32 (16.96) | 4.99 (14.17)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival was calculated as the time from the date of randomization to the date of death from any cause. Participants last known to be alive were censored at the last contact date.
Time Frame: From randomization until the end of study; median time on study was 9.64 months.
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 78 | 148
months | 10.9 [9.26 to 15.54] | 10.7 [8.54 to 12.35]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority; p = 0.5157, Log Rank; Log rank test stratified by the randomization stratification factors; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.81 to 1.53] — Based on a Cox proportional hazards model stratified by the randomized stratification factors. Hazard ratio < 1 favors denosumab

2. Secondary Outcome: Correlation of Tumor Tissue RANK Expression With Overall Survival
Description: To assess whether the treatment effect on overall survival was correlated with receptor activator of nuclear factor (NF)-κB (RANK) protein expression in tumor cells, RANK expression in archival tumor samples was measured using immunohistochemistry. The intensity of stain in the cytoplasm, membrane, and total was categorized as 0 (negative), 1+ (weak), 2+ (moderate) or 3+ (strong); All intensity is the sum of levels +1, +2 and +3. In addition, an H-score was calculated using the following formula: H-score=(percentage of cells of weak×1)+(percentage of cells of moderate×2)+(percentage of cells of strong×3). The maximum H-score was 300, corresponding to 100% of cells with strong intensity.
  The correlation between RANK expression level and OS was evaluated using a Cox proportional hazard models that included RANK expression level stratified by the randomization stratification factors in the corresponding treatment group.
Time Frame: From randomization until the data cut-off date of 29 July 2016; median time on study was 9.64 months.
Population: All randomized participants who had evaluable pre-treatment tumor RANK expression.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 64 | 123
hazard ratio
  Cytoplasm all intensity | 0.84 [0.65 to 1.09] | 1.00 [0.85 to 1.17]
  Membrane all intensity | 0.72 [0.51 to 1.01] | 0.92 [0.74 to 1.14]
  Total all intensity | 0.80 [0.62 to 1.03] | 1.00 [0.85 to 1.17]
  Cytoplasm H-score | 0.83 [0.65 to 1.07] | 1.00 [0.86 to 1.16]
  Membrane H-score | 0.72 [0.52 to 1.00] | 0.93 [0.77 to 1.13]
  Total H-score | 0.80 [0.62 to 1.02] | 1.00 [0.86 to 1.16]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; The interaction of RANK expression level measured in the cytoplasm (all intensity) and treatment effect was evaluated using a Cox proportional hazard model that included treatment group, RANK expression level and treatment-by-RANK expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.3759, Cox propotional hazard model
Statistical Analysis 2: Comparison: Placebo vs Denosumab; The interaction of RANK expression level measured in membranes (all intensity) and treatment effect was evaluated using a Cox proportional hazard model that included treatment group, RANK expression level and treatment-by-RANK expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.3666, Cox propotional hazard model
Statistical Analysis 3: Comparison: Placebo vs Denosumab; The interaction of RANK expression level total (cytoplasm + membranes; all intensity) and treatment effect was evaluated using a Cox proportional hazard model that included treatment group, RANK expression level and treatment-by-RANK expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.1917, Cox propotional hazard model
Statistical Analysis 4: Comparison: Placebo vs Denosumab; The interaction of RANK expression level measured in the cytoplasm (H-score) and treatment effect was evaluated using a Cox proportional hazard model that included treatment group, RANK expression level and treatment-by-RANK expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.3353, Cox propotional hazard model
Statistical Analysis 5: Comparison: Placebo vs Denosumab; The interaction of RANK expression level measured in membranes (H-score) and treatment effect was evaluated using a Cox proportional hazard model that included treatment group, RANK expression level and treatment-by-RANK expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.3179, Cox propotional hazard model
Statistical Analysis 6: Comparison: Placebo vs Denosumab; The interaction of RANK expression level total (cytoplasm + membranes; H-score) and treatment effect was evaluated using a Cox proportional hazard model that included treatment group, RANK expression level and treatment-by-RANK expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.1583, Cox propotional hazard model

3. Secondary Outcome: Correlation of Tumor Tissue RANK Ligand Expression With Overall Survival
Description: To assess whether the treatment effect on overall survival was correlated with RANK ligand (RANKL) protein expression in tumor cells, RANKL expression in archival tumor samples was measured using immunohistochemistry. The intensity of stain in the cytoplasm was categorized as 0 (negative), 1+ (weak), 2+ (moderate) or 3+ (strong); All intensity is the sum of levels +1, +2 and +3. In addition, an H-score was calculated using the following formula: H-score=(percentage of cells of weak×1)+(percentage of cells of moderate×2)+(percentage of cells of strong×3). The maximum H-score was 300, corresponding to 100% of cells with strong intensity.
  The correlation between RANKL expression level and OS was evaluated using a Cox proportional hazard models that included RANKL expression level stratified by the randomization stratification factors in the corresponding treatment group.
Time Frame: From randomization until the data cut-off date of 29 July 2016; median time on study was 9.64 months.
Population: All randomized participants who had evaluable pre-treatment tumor RANKL expression.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 65 | 121
hazard ratio
  Cytoplasm all intensity | 0.77 [0.63 to 0.95] | 0.93 [0.82 to 1.05]
  Cytoplasm H-score | 0.79 [0.66 to 0.95] | 0.93 [0.84 to 1.04]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; The interaction of RANKL expression level measured in the cytoplasm (all intensity) and treatment effect was evaluated using a Cox proportional hazard model that included treatment group, RANKL expression level and treatment-by-RANKL expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.3946, Cox propotional hazard model
Statistical Analysis 2: Comparison: Placebo vs Denosumab; The interaction of RANKL expression level measured in the cytoplasm (H-score) and treatment effect was evaluated using a Cox proportional hazard model that included treatment group, RANKL expression level and treatment-by-RANKL expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.3735, Cox propotional hazard model

4. Secondary Outcome: Objective Response Rate
Description: Objective response rate was defined as the percentage of participants with a complete response (CR) or partial response (PR) based on modified RECIST 1.1 achieved over the study duration.
  CR: Disappearance of all target and non target lesions, normalization of tumor marker levels and no new lesions.
  PR: At least a 30% decrease in the size of target lesions with no progression of non-target lesions and no new lesions, or, disappearance of target lesions with persistence of one or more non-target lesions and/or maintenance of tumor marker levels above normal limits and no new lesions.
  Participants who underwent surgical resection while on study were not evaluated for response after the surgery. Participants who did not meet the criteria for an objective response by the analysis cutoff date were considered non-responders.
Time Frame: From randomization until the data cut-off date of 29 July 2016; median time on study was 9.64 months.
Population: Randomized participants with at least one baseline measurable lesion per modified RECIST 1.1.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 76 | 144
percentage of participants | 43.4 | 36.8
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority or Other; p = 0.3491, Regression, Logistic; Logistic regression model adjusted for the randomization stratification factors; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.43 to 1.35] — Based on a logistic regression model adjusted for the randomization stratification factors; an odds ratio ≥ 1 favors denosumab

5. Secondary Outcome: Correlation of Tumor Tissue RANK Expression With Objective Response Rate
Description: To assess whether the treatment effect on objective response rate (ORR) based on RECIST 1.1 was correlated with RANK protein expression in tumor cells, RANK expression in archival tumor samples was measured using immunohistochemistry. The intensity of stain in the cytoplasm, membrane, and total was categorized as 0 (negative), 1+ (weak), 2+ (moderate) or 3+ (strong); All intensity is the sum of levels +1, +2 and +3. In addition, an H-score was calculated using the following formula: H-score=(percentage of cells of weak×1)+(percentage of cells of moderate×2)+(percentage of cells of strong×3). The maximum H-score was 300, corresponding to 100% of cells with strong intensity.
  The correlation between RANK expression level and ORR was evaluated within each treatment group using a logistical regression model that included RANK expression value as an independent variable and stratified by the randomization stratification factors. The odds ratio and 95% confidence interval are reported.
Time Frame: From randomization until the data cut-off date of 29 July 2016; median time on study was 9.64 months.
Population: All randomized participants with at least one baseline measurable lesion per modified RECIST 1.1 who had evaluable pre-treatment tumor RANK expression.
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 63 | 119
odds ratio
  Cytoplasm all intensity | 1.00 [0.67 to 1.50] | 0.88 [0.68 to 1.13]
  Membrane all intensity | 1.18 [0.74 to 1.89] | 0.82 [0.57 to 1.17]
  Total all intensity | 1.16 [0.78 to 1.71] | 0.88 [0.68 to 1.13]
  Cytoplasm H-score | 1.00 [0.69 to 1.47] | 0.87 [0.68 to 1.11]
  Membrane H-score | 1.14 [0.74 to 1.76] | 0.82 [0.59 to 1.14]
  Total H-score | 1.14 [0.79 to 1.65] | 0.87 [0.69 to 1.11]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; The interaction of RANK expression level measured in the cytoplasm (all intensity) and treatment effect was evaluated using a logistic regression model that included treatment group, RANK expression level and treatment-by-RANK expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.4760, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Denosumab; The interaction of RANK expression level measured in the membranes (all intensity) and treatment effect was evaluated using a logistic regression model that included treatment group, RANK expression level and treatment-by-RANK expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.2582, Regression, Logistic
Statistical Analysis 3: Comparison: Placebo vs Denosumab; The interaction of RANK expression level total (cytoplasm + membrane; all intensity) and treatment effect was evaluated using a logistic regression model that included treatment group, RANK expression level and treatment-by-RANK expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.2230, Regression, Logistic
Statistical Analysis 4: Comparison: Placebo vs Denosumab; The interaction of RANK expression level measured in the cytoplasm (H-score) and treatment effect was evaluated using a logistic regression model that included treatment group, RANK expression level and treatment-by-RANK expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.4329, Regression, Logistic
Statistical Analysis 5: Comparison: Placebo vs Denosumab; The interaction of RANK expression level measured in the membranes (H-score) and treatment effect was evaluated using a logistic regression model that included treatment group, RANK expression level and treatment-by-RANK expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.2620, Regression, Logistic
Statistical Analysis 6: Comparison: Placebo vs Denosumab; The interaction of RANK expression level total (cytoplasm + membrane; H-score) and treatment effect was evaluated using a logistic regression model that included treatment group, RANK expression level and treatment-by-RANK expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.2081, Regression, Logistic

6. Secondary Outcome: Correlation of Tumor Tissue RANKL Expression With Objective Response Rate
Description: To assess whether the treatment effect on objective response rate (ORR) based on RECIST 1.1 was correlated with RANKL protein expression in tumor cells, RANKL expression in archival tumor samples was measured using immunohistochemistry. The intensity of stain in the cytoplasm was categorized as 0 (negative), 1+ (weak), 2+ (moderate) or 3+ (strong); All intensity is the sum of levels +1, +2 and +3. In addition, an H-score was calculated using the following formula: H-score=(percentage of cells of weak×1)+(percentage of cells of moderate×2)+(percentage of cells of strong×3). The maximum H-score was 300, corresponding to 100% of cells with strong intensity.
  The correlation between RANKL expression level and ORR was evaluated within each treatment group using a logistical regression model that included RANKL expression value as an independent variable and stratified by the randomization stratification factors. The odds ratio and 95% confidence interval are reported.
Time Frame: From randomization until the data cut-off date of 29 July 2016; median time on study was 9.64 months.
Population: All randomized participants with at least one baseline measurable lesion per modified RECIST 1.1 who had evaluable pre-treatment tumor RANKL expression.
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 64 | 117
odds ratio
  Cytoplasm all intensity | 1.27 [0.88 to 1.83] | 1.10 [0.90 to 1.35]
  Cytoplasm H-score | 1.25 [0.91 to 1.72] | 1.09 [0.91 to 1.30]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; The interaction of RANKL expression level measured in the cytoplasm (all intensity) and treatment effect was evaluated using a logistic regression model that included treatment group, RANKL expression level and treatment-by-RANKL expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.4671, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Denosumab; The interaction of RANKL expression level measured in the cytoplasm (H-score) and treatment effect was evaluated using a logistic regression model that included treatment group, RANKL expression level and treatment-by-RANKL expression level interaction stratified by the randomization stratification factors; Test type: Superiority or Other; p = 0.4236, Regression, Logistic

7. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate was defined as the percentage of participants with an objective response (CR or PR) or stable disease (SD) or better for at least 16 weeks achieved over the study duration. If a participant underwent surgical resection while on study, the participant was not evaluated for response after the surgery. Participants who did not meet the criteria for clinical benefit by the analysis cutoff date were considered as non-responders.
Time Frame: From randomization until the data cut-off date of 29 July 2016; median time on study was 9.64 months.
Population: Randomized participants with at least one baseline measurable lesion per modified RECIST 1.1.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 76 | 144
percentage of participants | 53.9 | 47.9
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority or Other; p = 0.4654, Regression, Logistic; Logistic regression model adjusted for the randomization stratification factors; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.46 to 1.43] — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the time from randomization to the first observed disease progression per modified RECIST 1.1 criteria or death from any cause. Participants last known to be alive who did not experience disease progression were censored at their last imaging assessment date, last contact date if they were in the survival follow up phase, end of the study date, or the primary analysis cut-off date, whichever was first. If a participant underwent surgical resection while on study, the participant was censored at the last evaluable imaging assessment prior to the surgery.
Time Frame: From randomization until the data cut-off date of 29 July 2016; median time on study was 9.64 months.
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 78 | 148
months | 5.7 [4.37 to 7.16] | 5.2 [4.24 to 5.78]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority or Other; p = 0.7363, Log Rank; Log rank test stratified by the randomized stratification factors; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.78 to 1.43] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Serum Denosumab Trough Levels in Participants Who Received Q3W Dosing
Description: Serum samples were analyzed for denosumab using enzyme-linked immunosorbent assay (ELISA) following a validated procedure. The lower limit of quantification for the assay was 20 ng/mL.
Time Frame: Prior to dosing at day 8 and weeks 3, 6, 9, 12, 15, 18, 21 and 24.
Population: Randomized participants who received denosumab every 3 weeks with at least one valid denosumab concentration measurement.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Denosumab
Number analyzed (Participants) | 104
ng/mL
  Dose 2 - Day 8: number analyzed (Participants) | 63
  Dose 2 - Day 8 | 8590 (4080)
  Dose 3 - Week 3: number analyzed (Participants) | 17
  Dose 3 - Week 3 | 12200 (5710)
  Dose 4 - Week 6: number analyzed (Participants) | 46
  Dose 4 - Week 6 | 19700 (7350)
  Dose 5 - Week 9: number analyzed (Participants) | 56
  Dose 5 - Week 9 | 19600 (8270)
  Dose 6 - Week 12: number analyzed (Participants) | 51
  Dose 6 - Week 12 | 22800 (10400)
  Dose 7 - Week 15: number analyzed (Participants) | 46
  Dose 7 - Week 15 | 24300 (11500)
  Dose 8 - Week 18: number analyzed (Participants) | 40
  Dose 8 - Week 18 | 22700 (10600)
  Dose 9 - Week 21: number analyzed (Participants) | 31
  Dose 9 - Week 21 | 22100 (11200)
  Dose 10 - Week 24: number analyzed (Participants) | 28
  Dose 10 - Week 24 | 23300 (12700)

10. Secondary Outcome: Serum Denosumab Trough Levels in Participants Who Received Q4W Dosing
Description: as for outcome 9
Time Frame: Prior to dosing at day 8 and weeks 4, 8, 12, 16, 20 and 24
Population: Randomized participants who received denosumab every 4 weeks with at least one valid denosumab concentration measurement.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Denosumab
Number analyzed (Participants) | 8
ng/mL
  Dose 2 - Day 8: number analyzed (Participants) | 4
  Dose 2 - Day 8 | 8990 (2470)
  Dose 3 - Week 4: number analyzed (Participants) | 4
  Dose 3 - Week 4 | 10900 (3170)
  Dose 4 - Week 8: number analyzed (Participants) | 3
  Dose 4 - Week 8 | 15700 (6710)
  Dose 5 - Week 12: number analyzed (Participants) | 6
  Dose 5 - Week 12 | 14500 (4940)
  Dose 6 - Week 16: number analyzed (Participants) | 5
  Dose 6 - Week 16 | 13000 (4380)
  Dose 7 - Week 20: number analyzed (Participants) | 6
  Dose 7 - Week 20 | 15400 (5620)
  Dose 8 - Week 24: number analyzed (Participants) | 4
  Dose 8 - Week 24 | 15900 (7810)

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant. The event does not necessarily have a causal relationship with study treatment.
  A serious adverse event is defined as an AE that meets at least 1 of the following criteria
  * fatal
  * life threatening
  * requires in-patient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event Treatment-related AEs include only TEAEs for which the investigator indicated there was a reasonable possibility they may have been caused by study drug.
  Fatal adverse events include only deaths reported on the Adverse Event Case Report Form.
Time Frame: From first dose of study drug to the end of study date; the median (min, max) duration was 10.0 (0.2, 41.4) and 9.4 (0.2, 42.9) months for Placebo and Denosumab respectively.
Population: All randomized participants who received at least one dose of study drug (denosumab or placebo)
Measure: Number; unit: participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 76 | 145
participants
  All adverse events (AEs) | 76 | 144
  Serious adverse events | 68 | 129
  AEs leading to discontinuation of study drug | 6 | 20
  Fatal adverse events | 53 | 113
  Treatment-related adverse events (TRAEs) | 24 | 51
  Treatment-related serious adverse events | 0 | 6
  TRAEs leading to discontinuation of study drug | 0 | 7
  Treatment-related fatal adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug to the end of study date; the median (min, max) duration was 10.0 (0.2, 41.4) and 9.4 (0.2, 42.9) months for Placebo and Denosumab respectively.
Description: Data are included for all participants who received at least one dose of study drug.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Placebo: Participants received placebo matching to denosumab by subcutaneous injection once every 4 weeks (Q4W) plus one loading dose on study day 8 in addition to platinum-based standard chemotherapy. Participants may have received placebo as often as once every 3 weeks (Q3W) while receiving Q3W chemotherapy. Participants with bone metastases also received 4 mg zoledronic acid administered as an IV infusion Q4W or Q3W.
- Denosumab: Participants received 120 mg denosumab by subcutaneous injection once every 4 weeks plus one loading dose on study day 8 in addition to platinum-based standard chemotherapy. Participants may have received denosumab as often as Q3W while receiving Q3W chemotherapy. Participants with bone metastases also received placebo to zoledronic acid administered as an IV infusion Q4W or Q3W.
Arm/Group | Placebo | Denosumab
Serious Adverse Events (participants affected / at risk) | 68/76 | 129/145
Other Adverse Events (participants affected / at risk) | 71/76 | 139/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | Denosumab (N=145)
Anaemia (Blood and lymphatic system disorders) | 5 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 6
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 4
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 3 | 4
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Hereditary angioedema (Congenital, familial and genetic disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 6
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 4
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 4
Chills (General disorders) | 0 | 1
Condition aggravated (General disorders) | 1 | 1
Disease progression (General disorders) | 2 | 5
Fatigue (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 4 | 7
Infusion site extravasation (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 12
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2
Device related infection (Infections and infestations) | 1 | 1
Fungal infection (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis shigella (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Lung abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pleural infection (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 7 | 14
Respiratory tract infection (Infections and infestations) | 0 | 3
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 0 | 3
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1
Nutritional condition abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 3 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 4
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral lesion (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 9
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 10
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 19
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 14
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 12
Altered state of consciousness (Nervous system disorders) | 0 | 2
Brain oedema (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Consciousness fluctuating (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 2
Stroke in evolution (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Device issue (Product Issues) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 3
Delirium (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Renal haemorrhage (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Aortic thrombosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 0 | 1
Embolism venous (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 4
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | Denosumab (N=145)
Anaemia (Blood and lymphatic system disorders) | 38 | 60
Leukopenia (Blood and lymphatic system disorders) | 4 | 6
Neutropenia (Blood and lymphatic system disorders) | 15 | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 16
Dry eye (Eye disorders) | 4 | 2
Lacrimation increased (Eye disorders) | 3 | 9
Abdominal distension (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 13
Constipation (Gastrointestinal disorders) | 27 | 50
Diarrhoea (Gastrointestinal disorders) | 14 | 26
Dyspepsia (Gastrointestinal disorders) | 5 | 8
Dysphagia (Gastrointestinal disorders) | 6 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 6
Nausea (Gastrointestinal disorders) | 34 | 64
Stomatitis (Gastrointestinal disorders) | 6 | 7
Vomiting (Gastrointestinal disorders) | 14 | 35
Asthenia (General disorders) | 8 | 24
Fatigue (General disorders) | 33 | 67
Mucosal inflammation (General disorders) | 4 | 8
Oedema peripheral (General disorders) | 17 | 26
Pain (General disorders) | 7 | 10
Pyrexia (General disorders) | 9 | 23
Nasopharyngitis (Infections and infestations) | 5 | 3
Oral candidiasis (Infections and infestations) | 5 | 5
Pneumonia (Infections and infestations) | 2 | 10
Urinary tract infection (Infections and infestations) | 4 | 11
Fall (Injury, poisoning and procedural complications) | 5 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 3
Blood creatinine increased (Investigations) | 3 | 12
Platelet count decreased (Investigations) | 8 | 14
Weight decreased (Investigations) | 10 | 8
Decreased appetite (Metabolism and nutrition disorders) | 23 | 34
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 24
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 | 17
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 20
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 14
Dizziness (Nervous system disorders) | 7 | 20
Dysgeusia (Nervous system disorders) | 11 | 8
Headache (Nervous system disorders) | 8 | 24
Neuropathy peripheral (Nervous system disorders) | 9 | 5
Paraesthesia (Nervous system disorders) | 2 | 8
Anxiety (Psychiatric disorders) | 5 | 14
Depression (Psychiatric disorders) | 6 | 2
Insomnia (Psychiatric disorders) | 7 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 26
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 35
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 6
Rash (Skin and subcutaneous tissue disorders) | 8 | 18
Hypotension (Vascular disorders) | 5 | 4
Herpes zoster (Infections and infestations) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.